CLINICAL TRIAL: NCT01334216
Title: Using Computers to Assist in Parental Smoking Cessation in a Pediatric Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Stephen Downs, Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHICA_Smoking_Cessation_Study
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Results first posted 2017-03-14 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-08

CONDITIONS: Cigarette Smoking
Keywords: smoking; quitting; tobacco; Parental
MeSH Terms: conditions — Cigarette Smoking; Smoking

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CHICA Smoking Cessation Module (Active Comparator): This arm had the CHICA smoking cessation module turned on
  Interventions: Other: CHICA Smoking Cessation Module
- CHICA Placebo (Placebo Comparator): This arm had CHICA without the smoking cessation module
  Interventions: Other: CHICA Placebo

INTERVENTIONS:
Other: CHICA Smoking Cessation Module — The CHICA module helped to screen parents for smoking and assist them in quitting.
  Arms: CHICA Smoking Cessation Module
Other: CHICA Placebo — This was CHICA without the study module.
  Arms: CHICA Placebo

SUMMARY:
The CHICA system is a clinical decision support system that uses adaptive turnaround documents to provide point-of-care information to clinicians. The investigators will be studying whether it can help to support parents in their efforts to quit smoking.

DETAILED DESCRIPTION:
The CHICA system is a clinical decision support system that uses adaptive turnaround documents to provide point-of-care information to clinicians. The investigators will be studying in a randomized controlled trial whether it can help to support parents in their efforts to quit smoking.

ELIGIBILITY:
Inclusion Criteria:

Parent of child in our clinics who reported cigarette smoking

Exclusion Criteria:

Not smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2008-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Downs, MD, MS, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Children's Health Services Research, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CHICA Smoking Cessation Module | CHICA Placebo
Started | 168 | 194
Completed | 168 | 194
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CHICA Smoking Cessation Module | CHICA Placebo | Total
Number analyzed (Participants) | 168 | 194 | 362
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 168 | 194 | 362
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 106 | 194
  Male | 80 | 88 | 168
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 84 | 98 | 182
  White | 53 | 59 | 112
  Hispanic/Latino | 24 | 26 | 50
  Amer. Indian/Eskimo | 0 | 1 | 1
  Asian/Pacific Isl. | 5 | 6 | 11
  Other | 2 | 2 | 4
  Missing | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Parental Smoking Quit Rate
Description: This is the number of participants who quit smoking
Time Frame: one year
Measure: Count of Participants; unit: Participants
Arm/Group | CHICA Smoking Cessation Module | CHICA Placebo
Number analyzed (Participants) | 168 | 194
Participants | 31 | 20

ADVERSE EVENTS:
Time Frame: one year
Arm/Group | CHICA Smoking Cessation Module | CHICA Placebo
Serious Adverse Events (participants affected / at risk) | 0/168 | 0/194
Other Adverse Events (participants affected / at risk) | 0/168 | 0/194

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No